CLINICAL TRIAL: NCT02190292
Title: PANS - A Detailed Study of the Patients, Their Symptoms, Biomarkers and Treatment Offered in a Scandinavian Cohort
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Susanne Bejerot, Associate professor, Karolinska Institutet
Other Study IDs: 523-2011-3646_1
Record Dates: First submitted 2014-06-17; First posted 2014-07-15 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Obsessive-compulsive Disorder With Acute Onset; PANDAS; Pediatric Autoimmune Neuropsychiatric Disorders Associated With Streptococcal Infections; Pediatric Acute-onset Neuropsychiatric Syndrome (PANS); Childhood Acute Neuropsychiatric Symptoms (CANS); Obsessive-compulsive Disorder
MeSH Terms: conditions — Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal infections; Pediatric acute-onset neuropsychiatric syndrome; Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — blood (whole blood and serum)

GROUPS / COHORTS (3):
- PANS group: All current Swedish cases investigated with the Cunningham panel (approximately 150 individuals) will be invited to participate in the study. 50 of these will be re-assessed with the Cunningham panel.
- Psychiatric controls: 60 individuals with psychiatric disorder (eg. ADHD, autism spectrum disorder, psychosis, major depression, obsessive-compulsive disorder) will be recruited.
- Healthy controls: 25 age and sex matched children to the PANS group will be recruited.

SUMMARY:
Background: Obsessive-compulsive disorder (OCD) is considered one of the most debilitating of the psychiatric illnesses, yet much remains unclear regarding causes and cures. A diagnostic subgroup with acute onset of obsessive-compulsive symptoms (and sometimes tics or anorexia nervosa) possibly due to an autoimmune response, has been entitled Pediatric Acute onset Neuropsychiatric Syndrome (PANS). PANS is sometimes treated with immunomodulatory therapy or antibiotics, with a variable outcome. A diagnosis of PANS is supported by elevated levels of auto-antibodies and antibody-enzyme activity measured with the Cunningham panel, but the relationship between these biomarkers and the patients' symptoms remains unclear. A clinician rated symptom scale for PANS (the PANS scale) has been developed, but needs to be further evaluated regarding sensitivity and specificity.

Aims:

* To assess a Swedish cohort of patients diagnosed with PANS and compile their psychiatric health status, biomarkers, psychiatric symptoms, soft neurological signs and treatment outcomes in a systematic way
* To compare psychiatric health status, biomarkers and psychiatric, neurologic and motor symptoms in this PANS cohort with a control group of psychiatric patients and with healthy children.
* To evaluate the Cunningham panel as a diagnostic tool for PANS.
* To evaluate a clinician rated symptom scale (the PANS scale) as a diagnostic tool for PANS.

Method: Observational study Participants: Patients (n≈150) who have been tested with the Cunningham panel of PANS biomarkers in Sweden (or Swedish patients tested in Denmark) will be asked to participate.

Procedure: Assessment of current symptoms, psychiatric health, neurological and motor symptoms and possible biomarkers for PANS will be collected for all patients. Retrospective assessment through interview and medical records, including results from the first assessment with the Cunningham panel of PANS-biomarkers is made with all patients. 50 out of the total PANS cohort of 150 patients will be re-tested with the Cunningham panel. A control group consisting of psychiatric patients (n=60) and healthy children (n=25) will be examined with a similar test battery and signs and symptoms will be compared with the PANS group.

Significance:

Previous and current symptoms of PANS, levels of PANS biomarkers and treatment outcome will be investigated, thus knowledge regarding long-term outcome and evidence for the use of clinical assessment tools and biomarkers for diagnosing PANS will be gained.

DETAILED DESCRIPTION:
Data collected comprises:

Retrospective data

* Interview
* Medical records
* Five to Fifteen (FTF)
* Cunningham panel of PANS biomarkers result prior to inclusion (at time point 1)
* Change in Clinical Global Impression-Improvement (CGI-I) since the first assessment of the Cunningham panel

Current data

Current levels of Cunningham panel of PANS biomarkers

• Cunningham panel of PANS biomarkers at time point 2

Current neuropsychiatric status

* Psychiatric interview
* PANS symptom scale

Standardized assessment for children:

* Child behavior checklist (CBCL)
* The Autism spectrum Quotient: Children's version (AQ-Child)
* Brief Obsessive-Compulsive Scale (BOCS)
* Mini international Neuropsychiatric Interview - KID (M.I.N.I. KID)
* Five to Fifteen (FTF)

Standardized assessment for adults:

* Schizotypal Personality Disorder Questionnaire (SPQ)
* Liebowitz social anxiety scale (LSAS)
* The Autism spectrum Quotient (AQ)
* Adult ADHD Self-Report Scale (ASRS)
* Brown Attention-Deficit Disorder Scales (Brown ADD Scales)
* Quality of Life Inventory (QOLI)
* Brief obsessive-compulsive scale (BOCS)
* Mini international Neuropsychiatric Interview (M.I.N.I.)
* FTF retrospective data

Current soft neurological signs

* Alternating skips
* Romberg's balance test
* Diadochokinesia
* Involuntary finger movements

Current neuropsychological status

* Drawing exercises
* Writing exercises
* WAIS/WISC Block design
* WAIS/WISC Digit Span
* WAIS/WISC Letter Number Sequencing
* WAIS/WISC Digit Symbol Coding

Current biomarkers in blood/serum

* D8/17 antigen expression
* Human leukocyte antigen (HLA)
* C-reactive protein (CRP)
* T-cell activation
* Human proteome serum analysis

ELIGIBILITY:
Inclusion Criteria the PANS-group:

* Scandinavian patients assessed with the Cunningham panel through Wieslab, Lund, Sweden or Statens Serum Institut (SSI), Copenhagen, Denmark.

Exclusion Criteria PANS-group:

* intellectual disability, non-Swedish speaking

Inclusion Criteria Psychiatric Controls:

* diagnosed with a psychiatric disorder
* age <40 years

Exclusion Criteria Psychiatric Controls:

* intellectual disability, non-Swedish speaking

Inclusion Criteria Healthy Controls:

* age and sex matched to the PANS-group

Exclusion Criteria Healthy controls:

* intellectual disability, non-Swedish speaking

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive cases that have been assumed to have PANS and have been assessed with the Cunningham panel in Scandinavia.
Sampling Method: Probability Sample
Enrollment: 185 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Psychiatric health of individuals assessed with the Cunningham Panel of PANS-biomarkers | up to 4 years

SECONDARY OUTCOMES:
Sensitivity and Specificity of the Cuningham-Panel of PANS biomarkers as a diagnostic tool for PANS | up to 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Northern Stockholm psychiatry, Stockholm, Sverige, Sweden

REFERENCES:
- [Background] Bejerot S, Bruno K, Gerland G, Lindquist L, Nordin V, Pelling H, Humble MB. [Suspect PANDAS in children with acute neuropsychiatric symptoms. Infection behind the disease - long-term antibiotic therapy should be considered]. Lakartidningen. 2013 Oct 9-15;110(41):1803-6. No abstract available. Swedish. PMID 24187894
- [Background] Bernstein GA, Victor AM, Pipal AJ, Williams KA. Comparison of clinical characteristics of pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections and childhood obsessive-compulsive disorder. J Child Adolesc Psychopharmacol. 2010 Aug;20(4):333-40. doi: 10.1089/cap.2010.0034. PMID 20807071
- [Background] Brimberg L, Benhar I, Mascaro-Blanco A, Alvarez K, Lotan D, Winter C, Klein J, Moses AE, Somnier FE, Leckman JF, Swedo SE, Cunningham MW, Joel D. Behavioral, pharmacological, and immunological abnormalities after streptococcal exposure: a novel rat model of Sydenham chorea and related neuropsychiatric disorders. Neuropsychopharmacology. 2012 Aug;37(9):2076-87. doi: 10.1038/npp.2012.56. Epub 2012 Apr 25. PMID 22534626
- [Background] Demiroren K, Yavuz H, Cam L, Oran B, Karaaslan S, Demiroren S. Sydenham's chorea: a clinical follow-up of 65 patients. J Child Neurol. 2007 May;22(5):550-4. doi: 10.1177/0883073807302614. PMID 17690060
- [Background] Hachiya Y, Miyata R, Tanuma N, Hongou K, Tanaka K, Shimoda K, Kanda S, Hoshino A, Hanafusa Y, Kumada S, Kurihara E, Hayashi M. Autoimmune neurological disorders associated with group-A beta-hemolytic streptococcal infection. Brain Dev. 2013 Aug;35(7):670-4. doi: 10.1016/j.braindev.2012.10.003. Epub 2012 Nov 9. PMID 23142103
- [Background] Kirvan CA, Swedo SE, Heuser JS, Cunningham MW. Mimicry and autoantibody-mediated neuronal cell signaling in Sydenham chorea. Nat Med. 2003 Jul;9(7):914-20. doi: 10.1038/nm892. PMID 12819778
- [Background] Kirvan CA, Swedo SE, Snider LA, Cunningham MW. Antibody-mediated neuronal cell signaling in behavior and movement disorders. J Neuroimmunol. 2006 Oct;179(1-2):173-9. doi: 10.1016/j.jneuroim.2006.06.017. Epub 2006 Jul 27. PMID 16875742
- [Background] Kurlan R, Johnson D, Kaplan EL; Tourette Syndrome Study Group. Streptococcal infection and exacerbations of childhood tics and obsessive-compulsive symptoms: a prospective blinded cohort study. Pediatrics. 2008 Jun;121(6):1188-97. doi: 10.1542/peds.2007-2657. PMID 18519489
- [Background] Leckman JF, King RA, Gilbert DL, Coffey BJ, Singer HS, Dure LS 4th, Grantz H, Katsovich L, Lin H, Lombroso PJ, Kawikova I, Johnson DR, Kurlan RM, Kaplan EL. Streptococcal upper respiratory tract infections and exacerbations of tic and obsessive-compulsive symptoms: a prospective longitudinal study. J Am Acad Child Adolesc Psychiatry. 2011 Feb;50(2):108-118.e3. doi: 10.1016/j.jaac.2010.10.011. Epub 2010 Dec 31. PMID 21241948
- [Background] Leonard HL, Swedo SE. Paediatric autoimmune neuropsychiatric disorders associated with streptococcal infection (PANDAS). Int J Neuropsychopharmacol. 2001 Jun;4(2):191-8. doi: 10.1017/S1461145701002371. PMID 11466169
- [Background] Mabrouk AA, Eapen V. Challenges in the identification and treatment of PANDAS: a case series. J Trop Pediatr. 2009 Feb;55(1):46-8. doi: 10.1093/tropej/fmn039. Epub 2008 May 22. PMID 18499734
- [Background] Morris-Berry CM, Pollard M, Gao S, Thompson C; Tourette Syndrome Study Group; Singer HS. Anti-streptococcal, tubulin, and dopamine receptor 2 antibodies in children with PANDAS and Tourette syndrome: single-point and longitudinal assessments. J Neuroimmunol. 2013 Nov 15;264(1-2):106-13. doi: 10.1016/j.jneuroim.2013.09.010. Epub 2013 Sep 18. PMID 24080310
- [Background] Murphy TK, Goodman WK, Fudge MW, Williams RC Jr, Ayoub EM, Dalal M, Lewis MH, Zabriskie JB. B lymphocyte antigen D8/17: a peripheral marker for childhood-onset obsessive-compulsive disorder and Tourette's syndrome? Am J Psychiatry. 1997 Mar;154(3):402-7. doi: 10.1176/ajp.154.3.402. PMID 9054790
- [Background] Murphy TK, Kurlan R, Leckman J. The immunobiology of Tourette's disorder, pediatric autoimmune neuropsychiatric disorders associated with Streptococcus, and related disorders: a way forward. J Child Adolesc Psychopharmacol. 2010 Aug;20(4):317-31. doi: 10.1089/cap.2010.0043. PMID 20807070
- [Background] Murphy TK, Sajid M, Soto O, Shapira N, Edge P, Yang M, Lewis MH, Goodman WK. Detecting pediatric autoimmune neuropsychiatric disorders associated with streptococcus in children with obsessive-compulsive disorder and tics. Biol Psychiatry. 2004 Jan 1;55(1):61-8. doi: 10.1016/s0006-3223(03)00704-2. PMID 14706426
- [Background] Nicholson TR, Ferdinando S, Krishnaiah RB, Anhoury S, Lennox BR, Mataix-Cols D, Cleare A, Veale DM, Drummond LM, Fineberg NA, Church AJ, Giovannoni G, Heyman I. Prevalence of anti-basal ganglia antibodies in adult obsessive-compulsive disorder: cross-sectional study. Br J Psychiatry. 2012 May;200(5):381-6. doi: 10.1192/bjp.bp.111.092007. Epub 2012 Jan 26. PMID 22282431
- [Background] Perlmutter SJ, Leitman SF, Garvey MA, Hamburger S, Feldman E, Leonard HL, Swedo SE. Therapeutic plasma exchange and intravenous immunoglobulin for obsessive-compulsive disorder and tic disorders in childhood. Lancet. 1999 Oct 2;354(9185):1153-8. doi: 10.1016/S0140-6736(98)12297-3. PMID 10513708
- [Background] Singer HS, Gilbert DL, Wolf DS, Mink JW, Kurlan R. Moving from PANDAS to CANS. J Pediatr. 2012 May;160(5):725-31. doi: 10.1016/j.jpeds.2011.11.040. Epub 2011 Dec 22. No abstract available. PMID 22197466
- [Background] Swedo SE, Leonard HL, Garvey M, Mittleman B, Allen AJ, Perlmutter S, Lougee L, Dow S, Zamkoff J, Dubbert BK. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections: clinical description of the first 50 cases. Am J Psychiatry. 1998 Feb;155(2):264-71. doi: 10.1176/ajp.155.2.264. PMID 9464208
- [Background] Swedo SE, Leonard HL, Mittleman BB, Allen AJ, Rapoport JL, Dow SP, Kanter ME, Chapman F, Zabriskie J. Identification of children with pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections by a marker associated with rheumatic fever. Am J Psychiatry. 1997 Jan;154(1):110-2. doi: 10.1176/ajp.154.1.110. PMID 8988969
- [Background] Tan J, Smith CH, Goldman RD. Pediatric autoimmune neuropsychiatric disorders associated with streptococcal infections. Can Fam Physician. 2012 Sep;58(9):957-9. PMID 22972724
- [Background] Vincenzi B, O'Toole J, Lask B. PANDAS and anorexia nervosa--a spotters' guide: suggestions for medical assessment. Eur Eat Disord Rev. 2010 Mar;18(2):116-23. doi: 10.1002/erv.977. PMID 20148396
- [Derived] Hesselmark E, Bejerot S. Patient Satisfaction and Treatments Offered to Swedish Patients with Suspected Pediatric Acute-Onset Neuropsychiatric Syndrome and Pediatric Autoimmune Neuropsychiatric Disorders Associated with Streptococcal Infections. J Child Adolesc Psychopharmacol. 2019 Oct;29(8):634-641. doi: 10.1089/cap.2018.0141. Epub 2019 Apr 19. PMID 31009235